CLINICAL TRIAL: NCT05655156
Title: Post Market Clinical Follow-Up of OrthoPureXT for the Treatment of Multiligament Injured Knee: a Case Series
Brief Title: OrthoPureXT Multiligament PMCF Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tissue Regenix Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A03/0028/P01
Record Dates: First submitted 2022-11-16; First posted 2022-12-19 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-07

CONDITIONS: Multiligament Knee Injuries
Keywords: MLKI; PMCF; ACL PCL MCL LCL; IKDC; KOOS; Lysholm; Xenograft; MLKIs; Knee reconstruction; Knee injuries
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Intervention Model Description: Subjects with multiligament knee injuries will be evenly distributed across potential ligament reconstruction treatment options: PCL, ACL, MCL, LCL.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multiple Knee Ligament Injuries (Experimental): Sub-groups of n=7 incurring ligament reconstruction using OrthoPureXT in the following anatomical locations:
  * Posterior cruciate ligament (PCL)
  * Anterior cruciate ligament (ACL)
  * Posteromedial corner including the medial collateral ligament (MCL)
  * Posterolateral corner including the lateral collateral ligament (LCL)
  Interventions: Device: OrthoPure XT

INTERVENTIONS:
Device: OrthoPure XT — Indication: reconstruction of knee ligaments to restore knee function and stability
  The following device sizes are available for use in this indication:
  * Size 5
    - Multi-ligament reconstruction (recommended for extra-articular ligament reconstruction)
  * Size 6
    - Multi-ligament reconstruction (recommended for extra-articular ligament reconstruction)
  * Size 8
    * Primary ACL reconstruction where autograft tissue is not suitable
    * Revision ACL reconstruction
    * Multi-ligament reconstruction (recommended for extra-articular ligament reconstruction)
  * Size 10
    * Multi-ligament reconstruction (recommended for posterior cruciate ligament (PCL) reconstruction)

SUMMARY:
To monitor residual risks in the post-market phase and to ensure continued clinical evaluation of the device safety and performance to ensure that no new or unexpected risks arise when used during multi-ligament knee reconstructions.

DETAILED DESCRIPTION:
OrthoPureXT is an acellular, sterile, single use, xenograft (porcine) tissue scaffold that is manufactured using a proprietary decellularisation technology that renders the tissue substantially free from cells, leaving the porcine tissue biocompatible, and safe for implantation into the knee.

28 patients in total to be evenly distributed across potential ligament reconstruction treatment options (n=7 per sub-group) and resulting in a statistically relevant number per sub-group considering potential loss to follow up.

Sub-groups of n=7 incurring ligament reconstruction using OrthoPure XT in the following anatomical locations:

* Posterior cruciate ligament (PCL)
* Anterior cruciate ligament (ACL)
* Posteromedial corner including the medial collateral ligament (MCL)
* Posterolateral corner including the lateral collateral ligament (LCL)

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 years old or above.
* Adults suffering with multiple knee ligament injuries.
* Ability to communicate meaningfully with investigative staff, competence to give written informed consent; and willingness and ability to comply with entire study procedures including rehabilitation protocol.

Exclusion Criteria:

* Those unable to give consent.
* Those considered as conflicting variables by the investigator. This may include, but is not limited to:

  * Open trauma
  * Neurovascular emergencies
  * Compartment syndrome
  * Life threatening injury
* Those considered as physical barriers by the investigator, preventing physical or ethical collection of study data. This may include, but is not limited to:

  * Associated fractures that require external fixators
  * Local severe concomitant injuries
  * Injuries to other parts of the body associated with a high level of daily activity/intervention for the patient
* Those considered as a poor candidate for surgery by the investigator.
* If female and of child-bearing potential must not have a positive pregnancy test at Visit

  1 nor have a stated intention to become pregnant in the next 12 months.
* Those patients contraindicated for in the IFU, i.e.:

  * Showing signs of infection within 24 hours prior to surgery
  * Patients with known allergy, hypersensitivity, or religious objection to, implanted porcine material
  * Patients unable or unwilling to follow the post-operative care and rehabilitation programme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
A change from Baseline in IKDC | Baseline (30 days prior to surgery); 1, 3, 6 months after surgery (normal clinical follow-up); 12 and 24 months after surgery (long term follow-up)
  Assessment of knee stability via evaluation of IKDC score.

SECONDARY OUTCOMES:
A change from Baseline in Lysholm | Baseline (30 days prior to surgery); 1, 3 ,6 months after surgery (normal clinical follow-up); 12 and 24 months after surgery (long term follow-up)
  Assessment of knee stability via evaluation of Lysholm score.
A change from Baseline in KOOS | Baseline (30 days prior to surgery); 1, 3, 6 months after surgery (normal clinical follow-up); 12 and 24 months after surgery (long term follow-up)
  Assessment of knee stability via evaluation of KOOS.
A change from Baseline in Assessment of Laxity via Physical Examination | Baseline (30 days prior to surgery); 1, 3, 6 months after surgery (normal clinical follow-up); 12 and 24 months after surgery (long term follow-up)
  Physical assessment of passive movement focusing on the reconstructed ligament.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Stoke University Hospital, Stoke-on-Trent, United Kingdom

IPD SHARING:
Plan to Share IPD: No